CLINICAL TRIAL: NCT05902975
Title: Evaluation of the Antimicrobial Fiber Reinforced Composite Resin Space Maintainer Modified With Silver Nano Particles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Nada Mohamed Elsadany, Mohamed nada Mohamed elsadany, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Space maintainer
Record Dates: First submitted 2023-05-21; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Dental Caries in Children

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber reinforced composite space maintainer (Experimental): 12 children received fiber reinforced composite (FRC) space maintainer without silver nanoparticle.
  Interventions: Device: Fiber reinforced composite resin space maintainer
- Fiber reinforced space maintainer with silver nano particles (Experimental): 12 children received fiber reinforced composite (FRC) space maintainers modified with silver nanoparticles.
  Interventions: Device: Fiber reinforced composite resin space maintainer

INTERVENTIONS:
Device: Fiber reinforced composite resin space maintainer — Bonding of fiber reinforced with composite resin on primary second molar and primary canine under rubber dam isolation

SUMMARY:
Fiber reinforced composite resin space maintainer

DETAILED DESCRIPTION:
Evaluation of the antimicrobial fiber reinforced composite resin space maintainer modified by silver nano particles.

ELIGIBILITY:
Inclusion Criteria:

* Premature loss of primary molar.
* Presence of teeth on the mesial and distal sides of the extraction space.
* Normal primary molar relation.
* No root resorption of abutment teeth.
* Presence of a succedaneous tooth bud.
* Absence of pathology on the eruption track of the succedaneous tooth.
* The age will be ranged from 4 to 9 years.

Exclusion Criteria:

* Carious buccal and lingual surface of abutment teeth.
* Absence of teeth on the mesial and distal sides of the extraction.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2022-05-21 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of strepetoccous mutant and lactobacilli from sample of saliva | 6 month
  Streptococcus mutants : One loop (1/1000th ml of sample) was inoculated on the Mitis Salivarius (MSA)* agar with 0.2 U/ml bacitracin and sucrose (15% w/v) bacitracin. The plates were incubated aerobically ( 5% CO2) at 37°C for 48 h.(10) For determination of S. mutans count: After 48 h , colony characteristics were studied and the number of colony forming units of SM (CFU/ml) in saliva was determined manually .
  Lactobacilli : One loop (1/1000th ml of sample) was inoculated on the Rogosa **SL agar plate. The plates were incubated aerobically ( 5% CO2) at 37°C for 48 h.(11) For determination of lactobacilli count: After 48 h , colony characteristics were studied and the number of colony forming units of lactobacilli (CFU/ml) in saliva was determined manually

CONTACTS AND LOCATIONS:
Overall Officials: Alaa eldin Mahmoud Abdallah, Study Director — Associate professior; Hamdy Mahmoud Badereldin, Study Director — Lecture; Ahmed Akram Elawady, Study Director — Lecture
Locations (1):
- Alazhar university, Cairo, Egypt